CLINICAL TRIAL: NCT01576042
Title: Catheter Ablation for Ventricular Tachycardia in Patients With an Implantable Cardioverter Defibrillator (CALYPSO) PILOT TRIAL
Brief Title: Pilot Study of Catheter Ablation for Ventricular Tachycardia in Patients With an Implantable Cardioverter Defibrillator
Acronym: CALYPSO
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Main objectives of the study were met; consensus among investigators that continuing the study would not add new information beyond that already learned.
Sponsor: Duke University (Other)
Collaborators: Duke Clinical Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pro00033180; Pro00036518 (Other: Duke Site Protocol Number)
Record Dates: First submitted 2012-04-03; First posted 2012-04-12 (Estimated); Results first posted 2014-09-25 (Estimated); Last update posted 2014-10-16 (Estimated); Status verified 2014-09

CONDITIONS: Ventricular Tachycardia
Keywords: Ischemic heart disease; Implantable Cardioverter Defibrillator; Ventricular Tachycardia; Patient with Implantable Cardioverter Defibrillator (ICD)
MeSH Terms: conditions — Tachycardia, Ventricular; Myocardial Ischemia | interventions — Amiodarone; Sotalol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Catheter ablation (Other): The only ablation catheter that will be allowed in this study will be the Biosense Webster's NAVI-STAR Thermo-Cool catheter as it is the only catheter that has been approved by the FDA for sustained monomorphic VT due to prior myocardial infarction in adults
  Interventions: Device: Biosense Webster's NAVI-STAR Thermo-Cool
- Antiarrhythmic medication (Other): The choice of antiarrhythmic medications will comply with the ACC/AHA 2006 Guidelines for Management of Patients with Ventricular Arrhythmias and the Prevention of Sudden Cardiac Death
  Interventions: Drug: amiodarone; Drug: sotalol

INTERVENTIONS:
Drug: amiodarone — The dosage of antiarrhythmic medications will comply with the ACC/AHA 2006 Guidelines for Management of Patients with Ventricular Arrhythmias and the Prevention of Sudden Cardiac Death.
  Other Names: Cordarone
  Arms: Antiarrhythmic medication
Drug: sotalol — The choice and dosage of antiarrhythmic medications will comply with the ACC/AHA 2006 Guidelines for Management of Patients with Ventricular Arrhythmias and the Prevention of Sudden Cardiac Death.
  Other Names: Betapace; Betapace AF; Sotalex; Sotacor
  Arms: Antiarrhythmic medication
Device: Biosense Webster's NAVI-STAR Thermo-Cool — The only ablation catheter that will be allowed in this study will be the Biosense Webster's NAVI-STAR Thermo-Cool catheter as it is the only catheter that has been approved by the FDA for sustained monomorphic VT due to prior myocardial infarction in adults.
  Arms: Catheter ablation

SUMMARY:
The purpose of this pilot trial is to determine the feasibility of a large, multi-center randomized clinical trial aimed to test whether a treatment strategy of percutaneous catheter ablation of ventricular tachycardia (VT) is superior to state-of-the-art pharmacologic therapy at reducing all-cause mortality in patients with an implantable cardioverter defibrillator (ICD) who receive therapy for VT in the absence of any reversible cause.

DETAILED DESCRIPTION:
This study will be conducted at up to 8 sites and will randomize 50 patients over 1 year to a strategy of catheter ablation (n=25) vs. state-of-the-art pharmacologic therapy (n=25). To be considered for enrollment in this pilot trial, patients must be at least 18 years of age and must have an ICD for a primary or secondary prevention indication, have ≥ 1 documented ICD shock or ≥ 3 ATP therapies for VT in the absence of a reversible cause that in the opinion of the treating physician requires further therapy and be eligible for both catheter ablation and at least 1 antiarrhythmic medication. Patients will be followed at 3 and 6 months and their vital status will be determined via a phone call at 12 months. Data on the safety and efficacy of therapies used in the pilot study will be collected. Of particular interest are adverse events resulting from the catheter ablation procedure and major side effects from antiarrhythmic medications.

ELIGIBILITY:
Inclusion Criteria:

* Have an ICD with or without cardiac resynchronization therapy (i.e. CRT-D) for a primary or secondary prevention indication
* Have ischemic heart disease defined as the presence of wall motion abnormalities and documented coronary artery disease (one ≥ 70% stenosis in ≥ 1 major coronary artery)
* Have ≥ 1 documented ICD shock or ≥ 3 ATP therapies within 6 months before randomization for VT in the absence of a reversible cause that in the opinion of the treating physician requires further therapy. The VT has to be monomorphic and at a rate of ≤ 260 bpm.
* Be at least 18 years of age
* Be eligible for catheter ablation
* Have no history of intolerance or contraindication to at least 1 of the following antiarrhythmic medications: amiodarone, sotalol, and mexiletine.

Exclusion:

* Patients who in the opinion of the treating physician should not receive additional therapy
* More than 30 days of amiodarone treatment in the past 3 months unless the patient has been on ≤ 200 mgs of amiodarone daily for atrial arrhythmias or premature ventricular contractions (PVCs) and the patient is eligible for a higher dose of amiodarone
* Incessant VT that necessitates immediate treatment
* Reversible causes of VT including but not limited to ischemia, decompensated HF, and electrolyte disturbances
* The presence of a contraindication to catheter ablation of VT (including the presence of a mobile ventricular thrombus; an acute MI, coronary revascularization, or a stroke in the preceding 30 days; unstable angina or NYHA class IV HF; a mechanical valve; or inability to receive anticoagulation or antithrombotic therapy)
* Patients with non-ischemic cardiomyopathy
* Patients with hypertrophic obstructive, restrictive, or infiltrative cardiomyopathy
* Patients with acute myocarditis, congenital heart disease, valvular disease likely to require surgery in the next 1 year, and/or inoperable obstructive valvular disease
* Patients with a heart transplant or who are expected to undergo cardiac transplantation within 12 months
* Patients with a left ventricular assist device
* Patients who are already on antiarrhythmic drug therapy (other than beta-blockers) for VT (patients will not be excluded if they are receiving antiarrhythmic drug therapy for atrial arrhythmias or PVCs if they are eligible for additional drug therapy for VT).
* Heritable arrhythmias or increased risk for torsade de pointes with class III drugs
* End stage renal disease requiring dialysis
* Estimated life expectancy of <1 year from a non-cardiac cause
* Women who are pregnant or who have childbearing potential and are not using a reliable method of contraception
* Inability to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2012-05; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sana M Al-Khatib, MD, MHS, Principal Investigator — Duke University; William Stevenson, MD, Principal Investigator — Brigham and Women's Hospital
Locations (5):
- United States (5):
  - Johns Hopkins Hospital, Baltimore, Maryland
  - Duke University Medical Center, Durham, North Carolina
  - Ohio State University Medical Center, Columbus, Ohio
  - Penn State Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania

REFERENCES:
- [Background] Myerburg RJ, Kessler KM, Castellanos A. Sudden cardiac death: epidemiology, transient risk, and intervention assessment. Ann Intern Med. 1993 Dec 15;119(12):1187-97. doi: 10.7326/0003-4819-119-12-199312150-00006. PMID 8239250
- [Background] Gilman JK, Jalal S, Naccarelli GV. Predicting and preventing sudden death from cardiac causes. Circulation. 1994 Aug;90(2):1083-92. doi: 10.1161/01.cir.90.2.1083. PMID 7913885
- [Background] Zipes DP, Wellens HJ. Sudden cardiac death. Circulation. 1998 Nov 24;98(21):2334-51. doi: 10.1161/01.cir.98.21.2334. No abstract available. PMID 9826323
- [Background] Zheng ZJ, Croft JB, Giles WH, Mensah GA. Sudden cardiac death in the United States, 1989 to 1998. Circulation. 2001 Oct 30;104(18):2158-63. doi: 10.1161/hc4301.098254. PMID 11684624
- [Background] Antiarrhythmics versus Implantable Defibrillators (AVID) Investigators. A comparison of antiarrhythmic-drug therapy with implantable defibrillators in patients resuscitated from near-fatal ventricular arrhythmias. N Engl J Med. 1997 Nov 27;337(22):1576-83. doi: 10.1056/NEJM199711273372202. PMID 9411221
- [Background] Moss AJ, Zareba W, Hall WJ, Klein H, Wilber DJ, Cannom DS, Daubert JP, Higgins SL, Brown MW, Andrews ML; Multicenter Automatic Defibrillator Implantation Trial II Investigators. Prophylactic implantation of a defibrillator in patients with myocardial infarction and reduced ejection fraction. N Engl J Med. 2002 Mar 21;346(12):877-83. doi: 10.1056/NEJMoa013474. Epub 2002 Mar 19. PMID 11907286
- [Background] Kadish A, Dyer A, Daubert JP, Quigg R, Estes NA, Anderson KP, Calkins H, Hoch D, Goldberger J, Shalaby A, Sanders WE, Schaechter A, Levine JH; Defibrillators in Non-Ischemic Cardiomyopathy Treatment Evaluation (DEFINITE) Investigators. Prophylactic defibrillator implantation in patients with nonischemic dilated cardiomyopathy. N Engl J Med. 2004 May 20;350(21):2151-8. doi: 10.1056/NEJMoa033088. PMID 15152060
- [Background] Bardy GH, Lee KL, Mark DB, Poole JE, Packer DL, Boineau R, Domanski M, Troutman C, Anderson J, Johnson G, McNulty SE, Clapp-Channing N, Davidson-Ray LD, Fraulo ES, Fishbein DP, Luceri RM, Ip JH; Sudden Cardiac Death in Heart Failure Trial (SCD-HeFT) Investigators. Amiodarone or an implantable cardioverter-defibrillator for congestive heart failure. N Engl J Med. 2005 Jan 20;352(3):225-37. doi: 10.1056/NEJMoa043399. PMID 15659722
- [Background] Epstein AE, DiMarco JP, Ellenbogen KA, Estes NA 3rd, Freedman RA, Gettes LS, Gillinov AM, Gregoratos G, Hammill SC, Hayes DL, Hlatky MA, Newby LK, Page RL, Schoenfeld MH, Silka MJ, Stevenson LW, Sweeney MO, Smith SC Jr, Jacobs AK, Adams CD, Anderson JL, Buller CE, Creager MA, Ettinger SM, Faxon DP, Halperin JL, Hiratzka LF, Hunt SA, Krumholz HM, Kushner FG, Lytle BW, Nishimura RA, Ornato JP, Page RL, Riegel B, Tarkington LG, Yancy CW; American College of Cardiology/American Heart Association Task Force on Practice Guidelines (Writing Committee to Revise the ACC/AHA/NASPE 2002 Guideline Update for Implantation of Cardiac Pacemakers and Antiarrhythmia Devices); American Association for Thoracic Surgery; Society of Thoracic Surgeons. ACC/AHA/HRS 2008 Guidelines for Device-Based Therapy of Cardiac Rhythm Abnormalities: a report of the American College of Cardiology/American Heart Association Task Force on Practice Guidelines (Writing Committee to Revise the ACC/AHA/NASPE 2002 Guideline Update for Implantation of Cardiac Pacemakers and Antiarrhythmia Devices): developed in collaboration with the American Association for Thoracic Surgery and Society of Thoracic Surgeons. Circulation. 2008 May 27;117(21):e350-408. doi: 10.1161/CIRCUALTIONAHA.108.189742. Epub 2008 May 15. No abstract available. PMID 18483207
- [Background] Hammill SC, Stevenson LW, Kadish AH, Kremers MS, Heidenreich P, Lindsay BD, Mirro MJ, Radford MJ, Wang Y, Lang CM, Harder JC, Brindis RG. Review of the registry's first year, data collected, and future plans. Heart Rhythm. 2007 Sep;4(9):1260-3. doi: 10.1016/j.hrthm.2007.07.021. Epub 2007 Jul 25. No abstract available. PMID 17765637
- [Background] Hammill SC, Kremers MS, Stevenson LW, Kadish AH, Heidenreich PA, Lindsay BD, Mirro MJ, Radford MJ, Wang Y, Curtis JP, Lang CM, Harder JC, Brindis RG. Review of the Registry's second year, data collected, and plans to add lead and pediatric ICD procedures. Heart Rhythm. 2008 Sep;5(9):1359-63. doi: 10.1016/j.hrthm.2008.07.015. Epub 2008 Jul 22. No abstract available. PMID 18774117
- [Background] Hammill SC, Kremers MS, Kadish AH, Stevenson LW, Heidenreich PA, Lindsay BD, Mirro MJ, Radford MJ, McKay C, Wang Y, Lang CM, Pontzer K, Rumsfeld J, Phurrough SE, Curtis JP, Brindis RG. Review of the ICD Registry's third year, expansion to include lead data and pediatric ICD procedures, and role for measuring performance. Heart Rhythm. 2009 Sep;6(9):1397-401. doi: 10.1016/j.hrthm.2009.07.015. Epub 2009 Jul 16. No abstract available. PMID 19716099
- [Background] Hammill SC, Kremers MS, Stevenson LW, Heidenreich PA, Lang CM, Curtis JP, Wang Y, Berul CI, Kadish AH, Al-Khatib SM, Pina IL, Walsh MN, Mirro MJ, Lindsay BD, Reynolds MR, Pontzer K, Blum L, Masoudi F, Rumsfeld J, Brindis RG. Review of the registry's fourth year, incorporating lead data and pediatric ICD procedures, and use as a national performance measure. Heart Rhythm. 2010 Sep;7(9):1340-5. doi: 10.1016/j.hrthm.2010.07.015. Epub 2010 Jul 18. No abstract available. PMID 20647056
- [Background] Poole JE, Johnson GW, Hellkamp AS, Anderson J, Callans DJ, Raitt MH, Reddy RK, Marchlinski FE, Yee R, Guarnieri T, Talajic M, Wilber DJ, Fishbein DP, Packer DL, Mark DB, Lee KL, Bardy GH. Prognostic importance of defibrillator shocks in patients with heart failure. N Engl J Med. 2008 Sep 4;359(10):1009-17. doi: 10.1056/NEJMoa071098. PMID 18768944
- [Background] Sweeney MO, Sherfesee L, DeGroot PJ, Wathen MS, Wilkoff BL. Differences in effects of electrical therapy type for ventricular arrhythmias on mortality in implantable cardioverter-defibrillator patients. Heart Rhythm. 2010 Mar;7(3):353-60. doi: 10.1016/j.hrthm.2009.11.027. Epub 2009 Dec 2. PMID 20185109
- [Background] Noyes K, Corona E, Veazie P, Dick AW, Zhao H, Moss AJ. Examination of the effect of implantable cardioverter-defibrillators on health-related quality of life: based on results from the Multicenter Automatic Defibrillator Trial-II. Am J Cardiovasc Drugs. 2009;9(6):393-400. doi: 10.2165/11317980-000000000-00000. PMID 19929037
- [Background] Cardiac Arrhythmia Suppression Trial (CAST) Investigators. Preliminary report: effect of encainide and flecainide on mortality in a randomized trial of arrhythmia suppression after myocardial infarction. N Engl J Med. 1989 Aug 10;321(6):406-12. doi: 10.1056/NEJM198908103210629. PMID 2473403
- [Background] Echt DS, Liebson PR, Mitchell LB, Peters RW, Obias-Manno D, Barker AH, Arensberg D, Baker A, Friedman L, Greene HL, et al. Mortality and morbidity in patients receiving encainide, flecainide, or placebo. The Cardiac Arrhythmia Suppression Trial. N Engl J Med. 1991 Mar 21;324(12):781-8. doi: 10.1056/NEJM199103213241201. PMID 1900101
- [Background] Cardiac Arrhythmia Suppression Trial II Investigators. Effect of the antiarrhythmic agent moricizine on survival after myocardial infarction. N Engl J Med. 1992 Jul 23;327(4):227-33. doi: 10.1056/NEJM199207233270403. PMID 1377359
- [Background] Waldo AL, Camm AJ, deRuyter H, Friedman PL, MacNeil DJ, Pauls JF, Pitt B, Pratt CM, Schwartz PJ, Veltri EP. Effect of d-sotalol on mortality in patients with left ventricular dysfunction after recent and remote myocardial infarction. The SWORD Investigators. Survival With Oral d-Sotalol. Lancet. 1996 Jul 6;348(9019):7-12. doi: 10.1016/s0140-6736(96)02149-6. PMID 8691967
- [Background] Aliot EM, Stevenson WG, Almendral-Garrote JM, Bogun F, Calkins CH, Delacretaz E, Della Bella P, Hindricks G, Jais P, Josephson ME, Kautzner J, Kay GN, Kuck KH, Lerman BB, Marchlinski F, Reddy V, Schalij MJ, Schilling R, Soejima K, Wilber D; European Heart Rhythm Association (EHRA); Registered Branch of the European Society of Cardiology (ESC); Heart Rhythm Society (HRS); American College of Cardiology (ACC); American Heart Association (AHA). EHRA/HRS Expert Consensus on Catheter Ablation of Ventricular Arrhythmias: developed in a partnership with the European Heart Rhythm Association (EHRA), a Registered Branch of the European Society of Cardiology (ESC), and the Heart Rhythm Society (HRS); in collaboration with the American College of Cardiology (ACC) and the American Heart Association (AHA). Heart Rhythm. 2009 Jun;6(6):886-933. doi: 10.1016/j.hrthm.2009.04.030. No abstract available. PMID 19467519
- [Background] Grimm W, Flores BT, Marchlinski FE. Shock occurrence and survival in 241 patients with implantable cardioverter-defibrillator therapy. Circulation. 1993 Jun;87(6):1880-8. doi: 10.1161/01.cir.87.6.1880. PMID 8504500
- [Background] Exner DV, Pinski SL, Wyse DG, Renfroe EG, Follmann D, Gold M, Beckman KJ, Coromilas J, Lancaster S, Hallstrom AP; AVID Investigators. Antiarrhythmics Versus Implantable Defibrillators. Electrical storm presages nonsudden death: the antiarrhythmics versus implantable defibrillators (AVID) trial. Circulation. 2001 Apr 24;103(16):2066-71. doi: 10.1161/01.cir.103.16.2066. PMID 11319196
- [Background] Pacifico A, Hohnloser SH, Williams JH, Tao B, Saksena S, Henry PD, Prystowsky EN. Prevention of implantable-defibrillator shocks by treatment with sotalol. d,l-Sotalol Implantable Cardioverter-Defibrillator Study Group. N Engl J Med. 1999 Jun 17;340(24):1855-62. doi: 10.1056/NEJM199906173402402. PMID 10369848
- [Background] Kuhlkamp V, Mewis C, Mermi J, Bosch RF, Seipel L. Suppression of sustained ventricular tachyarrhythmias: a comparison of d,l-sotalol with no antiarrhythmic drug treatment. J Am Coll Cardiol. 1999 Jan;33(1):46-52. doi: 10.1016/s0735-1097(98)00521-x. PMID 9935007
- [Background] Seidl K, Hauer B, Schwick NG, Zahn R, Senges J. Comparison of metoprolol and sotalol in preventing ventricular tachyarrhythmias after the implantation of a cardioverter/defibrillator. Am J Cardiol. 1998 Sep 15;82(6):744-8. doi: 10.1016/s0002-9149(98)00478-0. PMID 9761084
- [Background] Connolly SJ, Dorian P, Roberts RS, Gent M, Bailin S, Fain ES, Thorpe K, Champagne J, Talajic M, Coutu B, Gronefeld GC, Hohnloser SH; Optimal Pharmacological Therapy in Cardioverter Defibrillator Patients (OPTIC) Investigators. Comparison of beta-blockers, amiodarone plus beta-blockers, or sotalol for prevention of shocks from implantable cardioverter defibrillators: the OPTIC Study: a randomized trial. JAMA. 2006 Jan 11;295(2):165-71. doi: 10.1001/jama.295.2.165. PMID 16403928
- [Background] Zipes DP, Camm AJ, Borggrefe M, Buxton AE, Chaitman B, Fromer M, Gregoratos G, Klein G, Moss AJ, Myerburg RJ, Priori SG, Quinones MA, Roden DM, Silka MJ, Tracy C, Smith SC Jr, Jacobs AK, Adams CD, Antman EM, Anderson JL, Hunt SA, Halperin JL, Nishimura R, Ornato JP, Page RL, Riegel B, Blanc JJ, Budaj A, Dean V, Deckers JW, Despres C, Dickstein K, Lekakis J, McGregor K, Metra M, Morais J, Osterspey A, Tamargo JL, Zamorano JL; American College of Cardiology/American Heart Association Task Force; European Society of Cardiology Committee for Practice Guidelines; European Heart Rhythm Association; Heart Rhythm Society. ACC/AHA/ESC 2006 Guidelines for Management of Patients With Ventricular Arrhythmias and the Prevention of Sudden Cardiac Death: a report of the American College of Cardiology/American Heart Association Task Force and the European Society of Cardiology Committee for Practice Guidelines (writing committee to develop Guidelines for Management of Patients With Ventricular Arrhythmias and the Prevention of Sudden Cardiac Death): developed in collaboration with the European Heart Rhythm Association and the Heart Rhythm Society. Circulation. 2006 Sep 5;114(10):e385-484. doi: 10.1161/CIRCULATIONAHA.106.178233. Epub 2006 Aug 25. No abstract available. PMID 16935995
- [Background] Julian DG, Camm AJ, Frangin G, Janse MJ, Munoz A, Schwartz PJ, Simon P. Randomised trial of effect of amiodarone on mortality in patients with left-ventricular dysfunction after recent myocardial infarction: EMIAT. European Myocardial Infarct Amiodarone Trial Investigators. Lancet. 1997 Mar 8;349(9053):667-74. doi: 10.1016/s0140-6736(96)09145-3. PMID 9078197
- [Background] Cairns JA, Connolly SJ, Roberts R, Gent M. Randomised trial of outcome after myocardial infarction in patients with frequent or repetitive ventricular premature depolarisations: CAMIAT. Canadian Amiodarone Myocardial Infarction Arrhythmia Trial Investigators. Lancet. 1997 Mar 8;349(9053):675-82. doi: 10.1016/s0140-6736(96)08171-8. PMID 9078198
- [Background] Singh SN, Fletcher RD, Fisher SG, Singh BN, Lewis HD, Deedwania PC, Massie BM, Colling C, Lazzeri D. Amiodarone in patients with congestive heart failure and asymptomatic ventricular arrhythmia. Survival Trial of Antiarrhythmic Therapy in Congestive Heart Failure. N Engl J Med. 1995 Jul 13;333(2):77-82. doi: 10.1056/NEJM199507133330201. PMID 7539890
- [Background] International mexiletine and placebo antiarrhythmic coronary trial: I. Report on arrhythmia and other findings. Impact Research Group. J Am Coll Cardiol. 1984 Dec;4(6):1148-63. doi: 10.1016/s0735-1097(84)80133-3. PMID 6209318
- [Background] Calkins H, Epstein A, Packer D, Arria AM, Hummel J, Gilligan DM, Trusso J, Carlson M, Luceri R, Kopelman H, Wilber D, Wharton JM, Stevenson W. Catheter ablation of ventricular tachycardia in patients with structural heart disease using cooled radiofrequency energy: results of a prospective multicenter study. Cooled RF Multi Center Investigators Group. J Am Coll Cardiol. 2000 Jun;35(7):1905-14. doi: 10.1016/s0735-1097(00)00615-x. PMID 10841242
- [Background] Reddy VY, Reynolds MR, Neuzil P, Richardson AW, Taborsky M, Jongnarangsin K, Kralovec S, Sediva L, Ruskin JN, Josephson ME. Prophylactic catheter ablation for the prevention of defibrillator therapy. N Engl J Med. 2007 Dec 27;357(26):2657-65. doi: 10.1056/NEJMoa065457. PMID 18160685
- [Background] Stevenson WG, Wilber DJ, Natale A, Jackman WM, Marchlinski FE, Talbert T, Gonzalez MD, Worley SJ, Daoud EG, Hwang C, Schuger C, Bump TE, Jazayeri M, Tomassoni GF, Kopelman HA, Soejima K, Nakagawa H; Multicenter Thermocool VT Ablation Trial Investigators. Irrigated radiofrequency catheter ablation guided by electroanatomic mapping for recurrent ventricular tachycardia after myocardial infarction: the multicenter thermocool ventricular tachycardia ablation trial. Circulation. 2008 Dec 16;118(25):2773-82. doi: 10.1161/CIRCULATIONAHA.108.788604. Epub 2008 Dec 8. PMID 19064682
- [Background] Kuck KH, Schaumann A, Eckardt L, Willems S, Ventura R, Delacretaz E, Pitschner HF, Kautzner J, Schumacher B, Hansen PS; VTACH study group. Catheter ablation of stable ventricular tachycardia before defibrillator implantation in patients with coronary heart disease (VTACH): a multicentre randomised controlled trial. Lancet. 2010 Jan 2;375(9708):31-40. doi: 10.1016/S0140-6736(09)61755-4. PMID 20109864

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Catheter Ablation | Antiarrhythmic Medication
Started | 13 | 14
Switched to the Other Arm | 5 | 1
Completed | 11 | 14
Not Completed | 2 | 0
Not completed — Physician Decision | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Catheter Ablation | Antiarrhythmic Medication | Total
Number analyzed (Participants) | 13 | 14 | 27
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 7 | 7 | 14
  >=65 years | 6 | 7 | 13
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 2 | 2
  Male | 13 | 12 | 25
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 4 | 6
  White | 11 | 10 | 21
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 13 | 14 | 27

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Completed Month 3 Follow-Up
Description: Records participants who completed Month 3 Follow-Up Visit
Time Frame: 3 months
Measure: Number; unit: participants
Arm/Group | Catheter Ablation | Antiarrhythmic Medication
Number analyzed (Participants) | 11 | 14
participants | 11 | 12

2. Secondary Outcome: Number of Participants Completed Month 6 Follow-Up
Description: Records participants who completed Month 6 Follow-Up Visit
Time Frame: 6 Months
Measure: Number; unit: participants
Arm/Group | Catheter Ablation | Antiarrhythmic Medication
Number analyzed (Participants) | 11 | 14
participants | 7 | 10

3. Secondary Outcome: Number of Participants Had at Least One of the Efficacy Outcome Measurement
Description: Records participants who had at least one of the efficacy outcome measurement (including death, hospitalization due to VT)
Time Frame: 6 Months
Measure: Number; unit: participants
Arm/Group | Catheter Ablation | Antiarrhythmic Medication
Number analyzed (Participants) | 11 | 14
participants | 11 | 14

4. Secondary Outcome: Cardiovascular Hospitalizations
Description: Records participants hospitalized for VT during the study
Time Frame: Baseline, 6 months
Measure: Number; unit: participants
Arm/Group | Catheter Ablation | Antiarrhythmic Medication
Number analyzed (Participants) | 11 | 14
participants | 5 | 7

5. Secondary Outcome: Number of Participants Remained on Randomized Treatment Assignment
Description: Records participants who only received study treatment as randomized during the entire study
Time Frame: 6 month
Measure: Number; unit: participants
Arm/Group | Catheter Ablation | Antiarrhythmic Medication
Number analyzed (Participants) | 11 | 14
participants | 6 | 13

6. Secondary Outcome: Number of Participants Switched to Other Arm
Description: Records participants who received study treatment as randomized and later switched to other treatment arm during the study
Time Frame: 6 months
Measure: Number; unit: participants
Arm/Group | Catheter Ablation | Antiarrhythmic Medication
Number analyzed (Participants) | 11 | 14
participants | 5 | 1

7. Secondary Outcome: Time to First Recurrent ICD Therapy for VT
Description: Days from the date of the first study treatment to the date of first ICD recurrent therapy for VT.
Time Frame: Baseline, 6 months
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Catheter Ablation | Antiarrhythmic Medication
Number analyzed (Participants) | 11 | 14
Days | 70.1 (38.09) | 78.7 (62.08)

8. Secondary Outcome: Number of Participants Received Treatment Assigned
Description: Records participants who received study randomized treatment during the study
Time Frame: 6 months
Measure: Number; unit: participants
Arm/Group | Catheter Ablation | Antiarrhythmic Medication
Number analyzed (Participants) | 11 | 14
participants | 11 | 14

ADVERSE EVENTS:
Time Frame: Adverse events related to the procedure or the use of antiarrhythmic medications was collected thru 6 months
Description: All Serious and non serious adverse events related to the procedure or the use of antiarrhythmic medications was collected thru 6 months. All have been reported in the results.
Arm/Group | Catheter Ablation | Antiarrhythmic Medication
Serious Adverse Events (participants affected / at risk) | 6/13 | 7/14
Other Adverse Events (participants affected / at risk) | 7/13 | 7/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Catheter Ablation (N=13) | Antiarrhythmic Medication (N=14)
Ventricular Tachycardia (Cardiac disorders) | 4 | 2
Hematoma (Vascular disorders) | 1 | 0
Cardiac Failure (Cardiac disorders) | 5 | 1
Renal Failure (Renal and urinary disorders) | 1 | 0
Ileus (Gastrointestinal disorders) | 1 | 0
Pneumonia (Infections and infestations) | 1 | 0
Device Malfunction (General disorders) | 2 | 0
Aortic Thrombosis (Vascular disorders) | 0 | 1
Lung Neoplasm Malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Chest Pain (General disorders) | 0 | 1
Myocardial Infarction (Cardiac disorders) | 0 | 1
Syncope (Nervous system disorders) | 0 | 1
Anemia (Blood and lymphatic system disorders) | 0 | 1
Diabetes Mellitus (Metabolism and nutrition disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Catheter Ablation (N=13) | Antiarrhythmic Medication (N=14)
Ventricular Tachycardia (Cardiac disorders) | 3 | 2
Cardiac Failure (Cardiac disorders) | 2 | 1
Myocardial Infarction (Cardiac disorders) | 0 | 1
Hematoma (Vascular disorders) | 2 | 0
Aortic Thrombosis (Vascular disorders) | 0 | 1
Hypotension (Vascular disorders) | 1 | 0
Ileus (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 0
Chest Pain (General disorders) | 0 | 1
Device Malfunction (General disorders) | 1 | 0
Syncope (Nervous system disorders) | 0 | 2
Anemia (Blood and lymphatic system disorders) | 0 | 1
Pneumonia (Infections and infestations) | 1 | 0
Diabetes Mellitus (Metabolism and nutrition disorders) | 0 | 1
Lung Neoplasm Malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Renal Failure (Renal and urinary disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No